CLINICAL TRIAL: NCT02790671
Title: An Open-Label, One-Sequence, Two-Period Study to Evaluate the Effects of Itraconazole on the Pharmacokinetics of DS-8500a in Healthy Subjects
Brief Title: A Study to Determine the Effects of Itraconazole on the Pharmacokinetics (PK) of DS-8500 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS8500-A-U109
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2016-08

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — firuglipel; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single study arm (Experimental): DS-8500a and itraconazole
  Interventions: Drug: DS-8500a; Drug: Itraconazole

INTERVENTIONS:
Drug: DS-8500a — DS-8500a 25mg tablet
Drug: Itraconazole — 200mg itraconazole

SUMMARY:
Study will assess the effects of itraconazole on the pharmacokinetic (PK) parameters of single-dose DS-8500a in healthy subjects. This is an open-label study in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 45 y of age, with a Body-Mass Index (BMI) of 18 kg/m2 to 30 kg/m2, inclusive, at Screening.
* Good health as determined by evaluations performed at Screening and during Enrollment on Day -1.
* Negative serum pregnancy test at Screening and a negative urine pregnancy test during Enrollment on Day -1 for all female subjects. Additionally, female subjects must be:

  * Surgically sterile (ie, bilateral tubal ligation or removal of both ovaries and/or uterus at least 6 mo prior to dosing)
  * Naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive mo prior to dosing, with a follicle stimulating hormone (FSH) level at Screening of ≥ 40 mIU/mL
  * Non-lactating
* Male subjects must agree to contraception (condom with spermicide) in addition to having their female partner (if of childbearing potential) use another form of contraception (eg, an intrauterine device, diaphragm with spermicide, oral contraceptive, injectables, or subdermal hormonal implant) from the first dose until 12 wk following last administration. Also, male subjects must not donate sperm during the study and afterwards for a period of 12 wk.
* Provided written informed consent prior to participating in the study. Able to understand and willing to comply with all the study requirements, and willing to allow the collection of all blood and urine specimens.
* Negative urine test for drugs of abuse (opiates, benzodiazepines, amphetamines, cannabinoids, cocaine, barbiturates, phencyclidine), cotinine, and alcohol at Screening and During Enrollment on Day -1.
* Willingness to abstain from grapefruit/grapefruit juice and Seville oranges 10 d before the first dose of study drug on Day 1 until the end of the study on Day 31.
* Willingness to refrain from consuming food or beverages containing caffeine/xanthine and alcohol 24 h prior to Enrollment on Day -1 until the end of the study on Day 31.

Exclusion Criteria:

* History or current evidence of clinically significant cardiac, hepatic, renal, pulmonary, endocrine/metabolic, neurologic, infectious, gastrointestinal (ie, any condition which may affect drug absorption), hematologic, or oncologic disease.
* Laboratory results (serum chemistry, hematology, and urinalysis) outside of the normal range and considered clinically significant in the opinion of the PI. Liver function (AST, ALT, bilirubin) test results must be below the ULN at Screening and during Enrollment on Day -1.
* A QTcF interval duration > 450 msec at Screening.
* Participation in a previous DS-8500a study, or dosing with itraconazole, within 6 mo prior to the first dose.
* Known sensitivity to product components of DS-8500a and/or itraconazole.
* Current participation in another investigational study or prior participation in an investigational study within the past 30 d prior to the first dose.
* Use of any prescription or over-the-counter (OTC) medications (systemic or topical), vitamins, or dietary/herbal supplements, including St John's Wort (hypericin), within 14 d prior to the first dose.
* Consumption of more than 28 units of alcohol per wk (males) or 14 units of alcohol per wk (females), where 1 unit of alcohol equals 1/2 pint of beer, 4 ounces of wine, or 1 ounce of spirits, or significant history of alcoholism or drug/chemical abuse within the last 2 y.
* Use of tobacco products or nicotine-containing products, including smoking cessation aids, such as gums or patches, within 6 mo prior to the first dose.
* Positive test result for HBsAg, HCV, or HIV antibody.
* Employment by the clinic.
* Familial relationship (spouse and/or first degree relative) with another study participant.
* Any other reason that, in the opinion of the PI, precludes subject participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
maximum concentration (Cmax) of DS-8500a | Day 1 to Day 6
  To assess the effects of itraconazole on the pharmacokinetic (PK) parameters of single-dose DS-8500a
time of maximum concentration (Tmax) of DS-8500a | Day 1 to Day 6
  To assess the effects of itraconazole on the pharmacokinetic (PK) parameters of single-dose DS-8500a
Area under the concentration curve (AUC) of DS-8500a | Day 1 to Day 6
  To assess the effects of itraconazole on the pharmacokinetic (PK) parameters of single-dose DS-8500a

SECONDARY OUTCOMES:
Number and severity of adverse events | Day 1 to Day 31
  To assess the the safety of DS-8500a
change in physical examination findings | Day 1 to Day 31
  To assess the the safety of DS-8500a
change in 12-lead electrocardiogram | Day 1 to Day 31
  To assess the the safety of DS-8500a
change in vital sign measurements | Day 1 to Day 31
  To assess the the safety of DS-8500a
change in clinical laboratory test results | Day 1 to Day 31
  To assess the the safety of DS-8500a

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/